CLINICAL TRIAL: NCT05547724
Title: Interest of Virtual Reality for the Management of Hospitalized Pregnant Patients at Risk of Preterm Delivery
Acronym: OREV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: departure of the principal investigator without replacement
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 87RI22_0027 (OREV)
Record Dates: First submitted 2022-09-10; First posted 2022-09-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: High Risk of Preterm Delivery
Keywords: virtual reality; anxiety; prematurity; pregnancy
MeSH Terms: conditions — Anxiety Disorders; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality (Experimental)
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: Virtual reality — Virtual reality visit of the birth room, cesarean and pediatric hospitalization department: neonatology and neonatal intensive care

SUMMARY:
Patients at high risk of preterm birth are hospitalized with an high stress for their child's future. In order to better prepare the patient to a possible preterm delivery we use to propose her a visit of the neonatology unit. However, as a result of their obstetrical condition and of the pediatric staff disponibility, this visit is not always possible. Virtual Reality (VR) is well known to provide an immersive experience while staying in a unique place. Our project is to propose a virtual visit of the delivery room, neonatology unit and intensive care unit to all hospitalized patients at risk of preterm delivery in order to prepare and decompress them.

DETAILED DESCRIPTION:
Most of the future parents are unprepared to outcomes of their premature child and the neonatology unit visit has a demonstrated anxiolytic effect on them (decrease of 6.7 points on the State Trait Anxiety Inventory-form Y scale (STAI-Y1)) unfortunately, as a result of their obstetrical condition and of the pediatric staff disponibility, the visit of the neonatology unit is not always possible in time.

Furthermore VR is known to be an immersive experience wich had already proved its comforting interest during delivery or to prepare patient to a planned caesarean.

In this study we propose to all hospitalized and high risk of delivery early patients a virtual visit of the neonatology unit from their sit in the calm space of their room. If the patient doesn't tolerate or has some VR contraindication : a virtual visit is possible on digital tablet. The visit is presented after the foetal lung maturation by 48h of Betamethasone. Patients complete a STAI-Y-A survey before and after the experience and a Simulator Sickness Questionnaire (SSQ) questionary to evaluate their tolerance. All medical informations can be found in the medical record.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient
* Patient with high risk of preterm delivery
* > 24 Week of Gestation (WG) et ≤ 34 WG
* Patient who received corticosteroids for fetal lung maturation in the previous 24h
* Patient > 18 years old

Exclusion Criteria:

* Patient no speak french
* no read french
* > 34 WG
* Guardianship, curatorship, or under the protection of a conservator
* Foetus vital prognosis engaged
* Medical contraindication to virtual reality: Epilepsy, bipolarity, severe motion sickness ( evaluated by the patient herself : history of nausea, sweat, emesis during car, boat or airplane transportation … +/- preventive therapy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-03-26 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Impact of a virtual reality | Day 1
  evaluation of the impact of a virtual reality visit on the anxiety of hospitalized patients with a risk of preterm delivery with the STAI-YA questionary

SECONDARY OUTCOMES:
Number of deliveries | Hours 12
  Number of deliveries in the 12 following hours VR.
Number of patients experiencing an increase in uterine contractions | Hours 12
  Number of patients experiencing an increase in uterine contractions in the 12 following hours VR.
Number of patients with rupture of membranes | Hours 12
  Number of patients with rupture of membranes obstetrical complications in the 12 following hours VR.
Evolution of Heart rate kinetics | Day 2
  evolution of heart rate kinetics during VR in beats per minute within 48 hours
% of patients with Arterial hypotension | Day 2
  Proportion in % of patients with arterial hypotension within 2 hours after VR in mmHg
% of patients with difficulty falling asleep | Day 2
  Proportion in % of patients with difficulty falling asleep the night after the visit, self-reported at the next day's medical visit.
Consumption of anxiolytics and analgesics | Day 2
  Variation in the use of anxiolytics and analgesics
% of patients wtihCybercinetosis | Hours 2
  Individual mean score and number and proportion of patients with an SSQ score > 38/48
% of patients wtih Visit interruption | Hours 2
  proportion in % of patients who interrupted the visit
% of patients wtih Visit on tablet | Hours 2
  Proportion in % of patients who completed the visit on a tablet
Average length of visit in VR | through study completion, a maximum of 18 weeks
  Average length of visit for each patient
% of patients wtih Renewal of the visit in VR | through study completion, a maximum of 18 weeks
  Proportion in % of patients wishing to repeat the visit
overall satisfaction | through study completion, a maximum 18 weeks
  Description of the patient's overall satisfaction of this study with Lickert's scale (Score between 0 unnecessary and 10 very useful)

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges Univesity Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No